CLINICAL TRIAL: NCT00749892
Title: A Phase II Exploratory Study of Pre-Operative Treatment With Erlotinib (Tarceva) in Muscle Invasive or Recurrent Transitional Cell Carcinoma Requiring Cystectomy
Brief Title: Erlotinib Hydrochloride in Treating Participants With Muscle Invasive or Recurrent Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0704; NCI-2018-01833 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007-0704 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Bladder Urothelial Carcinoma; Recurrent Renal Pelvis Urothelial Carcinoma; Recurrent Ureter Urothelial Carcinoma; Recurrent Urethral Urothelial Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0a Renal Pelvis Cancer AJCC v8; Stage 0a Ureter Cancer AJCC v8; Stage 0a Urethral Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage 0is Renal Pelvis Cancer AJCC v8; Stage 0is Ureter Cancer AJCC v8; Stage 0is Urethral Cancer AJCC v8; Stage II Bladder Cancer AJCC v8; Stage II Renal Pelvis Cancer AJCC v8; Stage II Ureter Cancer AJCC v8; Stage II Urethral Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Participants receive erlotinib hydrochloride PO QD for 3-5 weeks in the absence of disease progression or unacceptable toxicity. Within 24 hours of the last dose, participants undergo cystectomy.
  Interventions: Drug: Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva

SUMMARY:
This phase II trial studies how well erlotinib hydrochloride works in Treating participants with muscle invasive urothelial cancer or urothelial cancer that has come back. Drugs used in chemotherapy, such as erlotinib hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the response rate (ie: pT0 rate) of patients with urothelial cancer treated with erlotinib prior to cystectomy.

SECONDARY OBJECTIVES:

I. To estimate the 4-year disease-free survival of patients with urothelial cancer treated with erlotinib prior to cystectomy.

II. To measure epithelial-mesenchymal transition (EMT) markers (E-cadherin, HER4, PDGFR-beta, vimentin, fibronectin) in pre- and post-treatment biopsies and correlate expression patterns with the biological responses measured below.

III. To quantify target inhibition, antiproliferation (KI-67), and apoptosis (terminal deoxynucleotidyl transferase dUTP nick end labeling [TUNEL]) in biopsies obtained from patients before, during, and after therapy.

IV. Interrogate membrane (phosphorylated EGFR) and downstream receptor signaling pathways (ERKs, AKT/mTOR, GSK-3beta) to provide further insight into whether or not a given tumor displays a biological response.

V. To correlate the changes in Ki-67 expression with changes in angiogenesis and angiogenesis related gene expression utilizing fluorescent tissue staining techniques that we have developed in the laboratory (such as two-color TUNEL, phosphor-receptor, and microvessel density.) VI. To profile messenger ribonucleic acid (mRNA) expression in pre- and post-treatment biopsies using Affymetrix arrays and correlate the changes observed with EMT, growth arrest, and apoptosis.

VII. To quantify EGFR copy number and correlate with changes observed with EMT, growth arrest, and apoptosis.

OUTLINE:

Participants receive erlotinib hydrochloride orally (PO) once daily (QD) for 3-5 weeks in the absence of disease progression or unacceptable toxicity. Within 24 hours of the last dose, participants undergo cystectomy.

After completion of study treatment, participants are followed up every 6 months for 1 year, then annually for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of urothelial cancer. This includes bladder cancer, in addition to other tumors of the urothelial lining including renal pelvis, ureteral, and urethral cancer. This group may include any patient requiring cystectomy, including patients with recurrent or extensive superficial disease (cTa-T1N0M0), CIS (carcinoma in situ), or muscle invasive disease (cT2-3aN0M0), whose tumor could not be completely removed at transurethral resection
* Patients with the following high-risk features: Micropapillary features (more than focal on pathology); Small cell carcinoma; 3-dimensional (D) mass on exam under anesthesia (EUA); Lymphovascular invasion; Hydronephrosis (unless in the opinion of the treating physician, this is not due to tumor); High grade (grade 3) tumors of the ureter, renal pelvis, or urethra, or tumors in these areas with radiographic abnormality large enough to recognize as an abnormal mass by computed tomography (CT) or magnetic resonance imaging (MRI) imaging; Direct invasion of the prostatic stroma or the vaginal wall (ie: cT4a disease) should be offered neoadjuvant cytoreductive chemotherapy (ie: cisplatin-based). Patients refusing or who are not considered candidates for cytoreductive chemotherapy may be considered eligible. Dr. Siefker-Radtke will be the final arbiter in determining eligibility for the trial
* Please note that the presence of variant histologic subtypes is acceptable, except in the case for small cell variant which is traditionally treated with cytoreductive chemotherapy. Patients with small cell who refuse recommended cytoreductive chemotherapy may still be considered eligible
* Patients must have an evaluation in the department of urology, and be deemed an acceptable surgical candidate
* Patients must NOT have clinical evidence of metastatic disease by either CT or MRI of the abdomen and pelvis, and chest x-ray. In the absence of a bone scan, patients should be free of bone pain and have an alkaline phosphatase < 1.5 x upper limit of normal (ULN) of the upper limit of normal, or a normal bone fraction of alkaline phosphatase. If these features are present, patients should have a bone scan and this should be interpreted as showing no evidence of metastatic disease in order to be eligible
* Patients, 18 years and older, must either be not of child bearing potential or have a negative pregnancy test within 2 weeks of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
* Absolute neutrophil count (ANC) >= 1,000/ul
* Platelets >= 75,000/microliters
* Creatinine =< 2.0 x institutional upper limit of normal (ULN), or a creatinine clearance of > 30 ml/min as calculated by Cockroft-Gault or by 24-hour urine collection
* Bilirubin =< 2.5 x ULN
* Aspartate aminotransferase (AST) =< 5.0 x ULN
* Zubrod performance status (PS) =< 2
* Patients with second malignancies are eligible provided that the expected outcome from the second cancer is such that this will not interfere in the delivery of this therapy, or in doing cystectomy, and provided that the expectation of survival from any prior malignancy is reliably > 4 years

Exclusion Criteria:

* Acute hepatitis or known human immunodeficiency virus (HIV)
* Active or uncontrolled infection
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction =< 40%
* Prior therapy specifically and directly targeting the EGFR pathway
* Patients with interstitial lung disease
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s)
* Patients with metastatic or surgically unresectable disease are not eligible for this study. In addition, patients who do not agree to surgery are not eligible for this trial
* Patients who have received prior systemic chemotherapy or radiation therapy for urothelial cancer are not eligible. Any prior intravesical chemotherapy is allowed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 6/9/2008 and concluded on 12/19/2011 in the medical clinic. Diagnosis of invasive transitional cell carcinoma in the bladder, upper tract or urethra tumors were required for participants who were candidates for cystectomy to be considered. Participants with high-risk features were generally excluded.
Pre-assignment Details: Erlotinib treatment milestone: Three participants decided to not start the study medication.
Groups:
- Pre-surgical Erlotinib Treatment: Erlotinib 150 mg by mouth daily for 3 weeks followed by cystectomy within 24 hours of the last dose.
Period: Overall Study
Arm/Group | Pre-surgical Erlotinib Treatment
Started | 34
Completed | 31
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Participants were stagged clinically before treatment began. The T discribes the tumor size; the larger the number is the more advanced the disease. The N indicates the lymphpnode involvemnt; zero indicates that no lymph nodes were believed to be cancerous.
Arm/Group | Pre-surgical Erlotinib Treatment
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 68 [53 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34
Clinical Staging [Count of Participants; unit: Participants] — Participants were staged clinically before treatment began. The T describes the tumor size; the larger the number is the more advanced the disease. The N indicates the lymphnode involvement; zero indicates that no lymph nodes were believed to be cancerous. Population: Three particpants withdrew from study treatment.
  Participants
    cTaN0: number analyzed (Participants) | 31
    cTaN0 | 1
    cT1N0: number analyzed (Participants) | 31
    cT1N0 | 10
    cT2N0: number analyzed (Participants) | 31
    cT2N0 | 17
    cT3aN0: number analyzed (Participants) | 31
    cT3aN0 | 1
    cT3bN0: number analyzed (Participants) | 31
    cT3bN0 | 1
    cT4aN0: number analyzed (Participants) | 31
    cT4aN0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The response rate is the number of patients with urothelial cancer treated with erlotinib prior to cystectomy. The response is defined as the absence of residual cancer in the surgical removed tissue (i.e., pT0). A responder is defined as a participant with the pathological stage of pT0 meaning that there is no evidence of disease.
Time Frame: Determined at the time of surgery or cystectomy
Population: two participants did not take any eroltinib and three participants stopped erlotinib early due to intolerable side effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-surgical Erlotinib Treatment
Number analyzed (Participants) | 26
Participants
  Number of Responders | 8
  Number of Non Responders | 18

2. Secondary Outcome: Estimated 4-Year Disease-Free Survival
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Evaluated for 2 months once drug therapy started.
Description: Toxicities were measured at weekly visit while on therapy using the NCI CTCAE v3.0.
Arm/Group | Pre-surgical Erlotinib Treatment
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 19/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-surgical Erlotinib Treatment (N=31)
Rash (Skin and subcutaneous tissue disorders) | 2
Decreased Neutrophils/Grabulocytes (Blood and lymphatic system disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Fatigue (General disorders) | 1
Infection-wound (Infections and infestations) | 1
Decreased Leukocytes (Total WBD) (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-surgical Erlotinib Treatment (N=31)
Rash (Skin and subcutaneous tissue disorders) | 15
Diarrhea (Gastrointestinal disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 5
Decreased Neutrophils/Grabulocytes (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-03-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT00749892/Prot_SAP_000.pdf